CLINICAL TRIAL: NCT00228618
Title: Dietary Effects of Sulfur Amino Acid Depletion and Repletion on Glutathione and Cysteine Pools.
Brief Title: Dietary Effects of Sulfur Amino Acids
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Dean Jones, PhD Professor, Emory University
Other Study IDs: 1098-2003
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Healthy
Keywords: oxidative stress; amino acids; dietary requirements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine the level of sulfur amino acids in the diet that is needed to maintaining glutathione antioxidant status. This information could prove very useful in medicine because it could allow identification of an optimal diet for control of antioxidant levels. This diet could be used in conjunction with other therapies in order to prevent or delay oxidative stress and any diseases that may result from this. Total study participation will include a screening visit and a 14-day study period where dietary intake of sulfur amino acids will be controlled. We aim to enroll 12 normal subjects at Emory University Hospital.The primary hypothesis is that steady-state GSH/GSSG and CYS/CYSS redox in human plasma will become oxidized due to SAA intake at 0% of the RDA and reduced due to SAA intake at 3X the RDA.

DETAILED DESCRIPTION:
The long-term objectives of this research are to improve the definition of optimal human SAA intake. This will include defining Dietary Reference Intakes (DRI), estimated average requirement (EAR), and the upper limit (UL) of intake by improving the understanding of the physiologic and pathologic responses to variatiation in SAA intake. Using high-resolution 1H-NMR, we plan on developing comprehensive metabolic profiles that can indicate when SAA intake is inadequate.

The specific aims of the current protocol are:

1. To determine whether steady-state GSH/GSSG or Cys/CySS redox in human plasma is oxidized due to sulfur amino acid intake at 0% of the RDA.
2. To determine whether steady-state GSH/GSSG or Cys/CySS becomes more reducing during dietary sulfur amino acid repletion with SAA at 3X the RDA.
3. To determine whether low or high sulfur amino acid intakes induce primary and secondary metabolic effects detectable by high-resolution 1H-NMR.

B. BACKGROUND AND SIGNIFICANCE:

Sulfur amino acids are involved in central metabolic processes. The biologically useful sulfur is derived almost exclusively from the amino acids methionine and cysteine. Methionine (Met) is an essential amino acid and is metabolized in individuals by the transulfuration pathway to form cysteine (Cys) (1). In addition to use in the primary sequence of most proteins, both Met and Cys are required for other metabolic functions. Met is converted to S-adenosylmethionine, which is used for methylation reactions (2) for structural and functional modifications of proteins, RNA and DNA, as well as synthesis of phospholipids and signaling molecules. The carbon skeleton of Met is also used for biosynthesis of polyamines, which are required for cell division and cell growth (3). Cysteine is used for biosynthesis of glutathione (GSH), coenzyme A, taurine and sulfate (4). GSH functions in redox regulation (5) and detoxification of oxidants and reactive electrophiles (6). Coenzyme A is central to fatty acid metabolism and the citric acid cycle; taurine is utilized for bile acid synthesis and osmotic regulation (7); sulfate is used as a structural component of oligosaccharides (8), transport of steroid hormones (9) and detoxification of foreign compounds (10). Thus, there is a requirement for adequate sulfur amino acid intake that extends beyond the need for adequate amounts to maintain normal protein synthesis and turnover.

Sulfur amino acid intake in humans is variable and optimal SAA intake has not been adequately defined. The average American diet contains about 100 g of protein daily (4); the mean SAA intake is about 2.4 g (11). Daily intakes range from < 0.3 g to > 5 g (11). Most of the SAA is derived from animal protein, which constitutes about 2/3 of the total protein intake. The content of SAA in legumes and some types of nuts is about half of that in animal protein while most other plant-derived foods contain only 10-20% of the SAA found in an equivalent amount of animal protein. Because plant-derived foods are low in total protein, individuals who do not consume animal protein are at risk of SAA deficiency. Conversely, if excess SAA has associated health risks due to H2S or other toxic metabolites generated by colonic flora, individuals consuming diets high in animal protein would be at risk (12). Hence, Dietary Reference Intake values for SAA are needed as a foundation for improved dietary guidelines.

Differences in quantity and timing of SAA intake can result in substantial effects on Met, Cys and GSH homeostasis. Animal studies show that there is a diurnal variation in hepatic GSH in which the level increases following consumption of foods high in Cys and decreases in the post-absorptive period (16-17). The total amount of Cys present in GSH in the human body is about 3 g, roughly equal to the SAA requirement for 3 d (13) so that the Cys supply/utilization pattern can be considered in 4 phases. In the first phase, systemic Cys supply is from dietary Cys and metabolism of dietary Met. During this phase, excess Cys signals enhanced catabolism (18). Under post-absorptive conditions, probably for a period of about a day, systemic supply of Cys occurs principally from hepatic release of GSH (14). Under these conditions, Cys metabolism continues to support biosynthetic needs for taurine and sulfate. Although not explicitly established for humans, diurnal variation in hepatic GSH in mice ceases after 24 h of fasting so that systemic Cys supply probably enters a third phase after about 24 h. In this phase, an increased fraction of total systemic supply is likely to be derived from non-hepatic tissues (e.g., skeletal muscle; 15). Because sulfate and taurine production normally occurs in the intestines and liver (19), a decline in utilization of Cys for these functions is expected during this phase. A fourth phase appears likely to occur after about 3 days in which conservation of Met and Cys would be maximal.

In addition, detoxification of foreign compounds by conjugation with GSH, sulfate or taurine requires utilization of Cys. Such use can impose a substantial SAA demand; for instance, metabolism of 4 doses of maximum strength acetaminophen, i.e., 4 g daily, will consume the equivalent of up to 250 mg Cys for GSH conjugation and 640 mg Cys for sulfate conjugation (13). This amount is very similar to the RDA for SAA. Thus, the combination of dietary and environmental factors affecting SAA homeostasis and the complex metabolic effects that can result from variation in SAA homeostasis emphasize the need for better means to evaluate adequacy of SAA nutrition. This need is present for otherwise healthy individuals and is accentuated in acute or chronic illness and during convalescence and metabolic/nutritional stabilization during recovery from illness. The lower intake level was selected because it is similar to the lower intake levels estimated from food frequency analysis (11). This level could occur with a vegetarian diet with a poor selection of foods, but would not be as extreme as found with prolonged fasting or starvation. The upper SAA intake level was selected because 3X RDA is about 20% above the average intake of SAA in this country, thus representing a somewhat high but otherwise normal SAA intake.

High resolution 1H-NMR and mass spectrometry provides an approach to investigate complex metabolic effects of diet. Traditional methods to investigate dietary and nutritional components have relied upon isolation and purification of substances with specific biologic activities. However, the very large number of compounds in the diet, the multiple effects of individual compounds, the metabolic changes in the compounds that occur after consumption and the complex interactions of the compounds limit the ability to unravel complex effects such as those due to variation in SAA intake during health, illness and recovery from illness.

Available high resolution metabolic analysis (21) such as 1H-NMR and mass spectrometry (MS) combined with bioinformatic tools provides a way to identify and establish a pattern of metabolic changes attributed to SAA deficiency and excess. We believe that if the environment is controlled and a dietary change (e.g. different level of SAA intake) is induced in an individual, observed metabolic changes can be ascribed to the dietary change. High resolution 1H-NMR and MS are well suited for investigating changes in body fluid composition because a large number of metabolites are present in body fluids, many metabolites can be detected simultaneously and these metabolites can be analyzed and quantified with minimal or no sample preparation. Examples are available from the studies of Nicholson and coworkers.

The use of multivariate statistical analysis of NMR data to evaluate metabolic responses of living systems is under development for toxicologic screening of pharmacologic compounds (24). The principles for detection of diet-related effects on health are the same as for the toxicologic use; in effect, nutritional deficiencies, excesses or intolerances can be viewed as toxicologic responses that are expressed in the metabolic profile. Thus, we believe that the information-rich character of the NMR spectra with MS data can provide a powerful approach to investigate both direct and indirect effects of nutritional variation in SAA intake. Given the fundamental roles of SAA metabolites in cell growth regulation, digestion, detoxification, antioxidant defense and hormonal signaling, and the potential risks of excess SAA intake, metabolic profiling by NMR could provide a useful approach to define optimum SAA intake and, in the future, to diagnose and treat SAA malnutrition.

Considerable information is available concerning the assignment of NMR spectra of urine and plasma (e.g., Ref 22-24, 38-39); this information will provide a useful guide to possible metabolites which could vary as a function of SAA intake. 2-D NMR and other techniques are available for peak identification. However, the goals of this project do not require identification of which chemical species change, only whether changes at specific frequencies can be attributed to variation in SAA intake.

Significance. The sulfur amino acids, Met and Cys, are highly variable in human foods and there are risks associated with both deficiency and excess. Both are required for physiologic processes in addition to maintenance of protein synthesis and nitrogen balance, and, in principle, excess of either could lead to generation of toxic sulfur metabolites in the colon. The present study will test 2 novel approaches to define dietary sulfur amino acid needs (i.e., plasma redox and metabolic analyses by NMR and MS). The results are expected to establish the feasibility of using these approaches for improved definition of Dietary Reference Intake values for these important nutrients.

ELIGIBILITY:
Inclusion Criteria:

* within 10% of ideal body weight

Exclusion Criteria:

* smoker
* illness

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2005-01; Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean P Jones, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States